CLINICAL TRIAL: NCT04416555
Title: Virtual Reality Distraction for Reduction in Acute Postoperative Pain
Brief Title: Virtual Reality Distraction for Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-769; R44DA049640 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: parallel assignment (one arm will receive the full immersive virtual reality experience and the other arm will receive a static presentation in the same device)
Who Masked: Participant, Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VR googles using exposure sham program (Placebo Comparator): The study groups will receive VR googles and the sham program
  Interventions: Device: Placebo comparator: VR googles and the non reality experience
- VR googles and the real VR program experience. (Active Comparator): The study group will receive the VR googles and the real VR program experience.
  Interventions: Device: Active Comparator: VR googles and the real VR program to enter act with and experience

INTERVENTIONS:
Device: Placebo comparator: VR googles and the non reality experience — parallel assignment (this arm will receive a static presentation in the same device)
  Arms: VR googles using exposure sham program
Device: Active Comparator: VR googles and the real VR program to enter act with and experience — Parallel assignment (this arm will receive the full immersive virtual reality experience
  Arms: VR googles and the real VR program experience.

SUMMARY:
Using a randomized controlled design, the investigators goal is to estimate the effect of VR on postoperative analgesia and opioid consumption.

DETAILED DESCRIPTION:
Specifically, the investigators propose to test the primary hypothesis that the use of AppliedVR software in Pico G2 4K headsets decreases acute postoperative pain scores (with a 1 point difference considered clinically important) compared to sham treatment on a 0-10 scale 15 minutes after each use in the first 48 hours after surgery or hospital discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Physical Status 1-3;
* Scheduled for elective, primary total hip arthroplasty;
* Anticipated hospitalization of at least 1 night;
* Expected to require parenteral opioids for postoperative pain;
* Able to use IV PCA systems.

Exclusion criteria:

* History of chronic pain or care by a pain management specialist;
* Use of more than 30 mg/day of oral oxycodone (or equivalent);
* Greater than 12 weeks of current and continued opioid use;
* History of seizures, epilepsy, motion sickness, stroke, dementia;
* Non-English speaking;
* Women who are pregnant or breastfeeding;
* History of substance use disorder.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabry Ayad, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Araujo-Duran J, Kopac O, Montalvo Campana M, Bakal O, Sessler DI, Hofstra RL, Shah K, Turan A, Ayad S. Virtual Reality Distraction for Reducing Acute Postoperative Pain After Hip Arthroplasty: A Randomized Trial. Anesth Analg. 2024 Apr 1;138(4):751-759. doi: 10.1213/ANE.0000000000006642. Epub 2023 Sep 6. PMID 37678233

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality (VR) Headset With the Real VR Program Experience: The study group will receive the VR headset and the real VR program experience.
- VR Headset Using Sham 2D Programs: The study groups will receive VR headset and sham, two-dimensional programs
Period: Overall Study
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Started | 55 | 58
Completed | 55 | 55
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: 113 patients were enrolled. 3 patients withdrew and requested to have their data excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 63 (9) | 64 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 26 | 29 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 49 | 98
  Black | 4 | 3 | 7
  Multiracial | 1 | 2 | 3
  Unavailable/Declined | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (6) | 32 (7) | 31.5 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (Numerical Rating Scale)
Description: The primary outcome was post-intervention pain score, adjusted for the corresponding pre-intervention pain score. Pain scores were measured by the Numerical Rating Scale which ranges from 0 (lowest pain) to 10 (highest pain) We targeted 3 interventions per day for each patient, and thus, correspondingly 3 pre-post pain measurements per day. The reported value is the least squares mean calculated using a mixed model for repeated measures.
Time Frame: From the end of surgery until 48 hours after surgery or discharge, whichever comes first
Population: 113 patients were enrolled. 3 withdrew and requested to have their data excluded. 4 patients had missing data for the primary outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Number analyzed (Participants) | 52 | 54
score on a scale | 3.4 (0.3) | 3.5 (0.2)
Statistical Analysis 1: Comparison: Virtual Reality (VR) Headset With the Real VR Program Experience vs VR Headset Using Sham 2D Programs; Test type: Superiority; p = 0.391, Mixed Models Analysis

2. Secondary Outcome: Total Opioid Consumption
Description: The investigators measured total opioid consumption converted to morphine milligram equivalents (MME).
Time Frame: End of surgery to 72 hours after surgery.
Population: 113 patients were enrolled. 3 patients withdrew and requested to have their data excluded. And 3 other patients had missing data for this outcome.
Measure: Geometric Least Squares Mean (Standard Error); unit: morphine milligrams equivalent
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Number analyzed (Participants) | 52 | 55
morphine milligrams equivalent | 6.8 (3.4) | 5.7 (2.6)
Statistical Analysis 1: Comparison: Virtual Reality (VR) Headset With the Real VR Program Experience vs VR Headset Using Sham 2D Programs; Test type: Superiority; p = 0.608, Regression, Linear

3. Secondary Outcome: Time Weighted Average Pain Score
Description: Pain scores collected by nursing staff every 4 hours during the first 48 hours after surgery. Pain scores were measured by the Numerical Rating Scale which ranges from 0 (lowest pain) to 10 (highest pain). The reported value is the least squares mean calculated using a mixed model for repeated measures.
Time Frame: End of surgery to 48 hours after surgery
Population: 113 patients were enrolled. 3 patients withdrew and requested to have their data excluded. And 5 other patients had missing data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Number analyzed (Participants) | 52 | 53
units on a scale | 4.3 (0.6) | 4.4 (0.6)
Statistical Analysis 1: Comparison: Virtual Reality (VR) Headset With the Real VR Program Experience vs VR Headset Using Sham 2D Programs; Test type: Superiority; p = 0.768, Mixed Models Analysis

4. Secondary Outcome: Perception of Video System Usability
Description: Patient's perception of video system usability was assessed using a validated questionnaire (System Usability Scale). The System Usability Scale is scored from 0 to 100 and higher scores are related with devices that are easier to use.
Time Frame: Once between last intervention time and hospital discharge (up to 8 days after end of surgery)
Population: 113 patients were enrolled. 3 patients withdrew and requested to have their data excluded. Five patients had missing data for this outcome due to being lost to follow up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Number analyzed (Participants) | 52 | 53
score on a scale | 75 [70 to 83] | 70 [65 to 83]
Statistical Analysis 1: Comparison: Virtual Reality (VR) Headset With the Real VR Program Experience vs VR Headset Using Sham 2D Programs; Test type: Superiority; p = 0.244, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Post Discharge Analgesia.
Description: Pain Outcomes Questionnaire Short Form, which evaluates five domains (pain, mobility, activities of daily living, vitality, negative affect and fear). The Pain Outcomes Questionnaire Short Form is scored from 0 to 190 and higher scores are related with worst pain outcomes.
Time Frame: One week (7 days) after hospital discharge
Population: 113 patients were enrolled. 3 patients withdrew and requested to have their data excluded. Nine patients had missing data for this outcome due to being lost to follow up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
Number analyzed (Participants) | 49 | 52
score on a scale | 67 [47 to 93] | 58 [40 to 87]
Statistical Analysis 1: Comparison: Virtual Reality (VR) Headset With the Real VR Program Experience vs VR Headset Using Sham 2D Programs; Test type: Superiority; p = 0.191, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: End of surgery up to 48 hours after surgery or discharge, whichever came first.
Arm/Group | Virtual Reality (VR) Headset With the Real VR Program Experience | VR Headset Using Sham 2D Programs
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT04416555/Prot_SAP_000.pdf